CLINICAL TRIAL: NCT00779155
Title: A Double-blind, Sham-stimulation Controlled Study of the Application of Magnetic Fields Using the Jacobson Resonator for the Treatment of Parkinson's Disease.
Brief Title: Study of Magnetic Fields for Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: pico-tesla Magnetic Therapies, LLC, pico-tesla Magnetic Therapies, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PD pilot 2
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inactive Resonator Therapy (Placebo Comparator): Inactive magnetic resonance therapy
  Interventions: Device: The Resonator control
- Active Resonator Therapy (Active Comparator): active magnetic resonance therapy
  Interventions: Device: The Resonator

INTERVENTIONS:
Device: The Resonator — active magnetic field therapy
  Arms: Active Resonator Therapy
Device: The Resonator control — inactive magnetic field therapy with placebo fields
  Arms: Inactive Resonator Therapy

SUMMARY:
The purpose of this study is to determine if low level magnetic fields may help to relieve symptoms of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD with motor fluctuations of at least 3-4 hours daily., Subject on levodopa, subject is ambulatory, maintain regular med schedule, willing and able to abstain from new PD treatments, Able to demonstrate correct completion of PD diaries, non-demented, adequate contraceptive measures, capable of giving full written consent.

Exclusion Criteria:

* any factors that will prevent subject from completing full course of therapy with the resonator, any factors preventing subject from attending clinic in the "off" state, atypical parkinsonism, no active brain tumors, strokes, hydrocephalus, any other neurologic or non-neurologic disorder which might affect the symptomatic expression of pts. parkinsonism, suffers from chronic pain, no meds that may produce parkinsonism, no psychiatric disturbance, Epilepsy, HIV, Cancer, History of ECT, Diabetic Neuropathy, Uncontrolled HTN, Advanced Pulmonary Disease, Known heart conditions such as cardiac arrythmias, previous PD surgical interventions, prosthetics comprised of ferrous metals, pacemakers, DBS, Uncontrolled, unstable or untreated medical illnesses, Consumption of more than 21 alcoholic drinks per week, Pregnant, breast feeding, developmental disability

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- pico-tesla Magnetic Therapies, Littleton, Colorado, United States

REFERENCES:
- [Result] O. Klepitskaya, R. Kumar, Efficacy and Safety of Low Level Electromagnetic Fields Treatment in Parkinson's Disease. Movement Disorders; Vol. 23, No. 11, 2008, pp. 1628-1637

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactive Resonator Device: inactive magnetic fields with placebo fields
- Active Resonator Device: Active pico-tesla magnetic fields
Period: Overall Study
Arm/Group | Inactive Resonator Device | Active Resonator Device
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactive Resonator Device | Active Resonator Device | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Study End Point in the Combined Scores From the UPDRS Subscale II and III Recorded in the Subjects "on" State.
Description: The UPDRS is used to measure different aspects of Parkinson's Disease (PD). The UPDRS subscale II assesses how PD affects a person's daily life, with scores ranging from 0-52, with 52 representing greatest severity. The UPDRS subscale III assesses how PD affects how a person moves about, with scores ranging from 0-108, with 108 representing greatest severity. The combination of these 2 scores is used in clinical trials and in clinical practice to get a good overall idea of how PD affects a person's life. Combined score ranges from 0-160, with 160 being greatest severity.
Time Frame: Baseline and 8 weeks
Population: Analysis was by intention to treat and all enrolled subjects completed the entire protocol.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Inactive Resonator Device | Active Resonator Device
Number analyzed (Participants) | 6 | 6
scores on a scale | -1 (.5) | -5 (1.2)

ADVERSE EVENTS:
Arm/Group | Inactive Resonator Device | Active Resonator Device
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes